CLINICAL TRIAL: NCT06527625
Title: Cultural Arts for Reducing Depressive Symptoms and Age-related Self-stigma in Older People: a Randomised Waitlist Controlled Trial
Brief Title: Cultural Arts Programme for Older Chinese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, LIU Tianyin Bridget, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20240227002
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Depressive Symptoms; Ageism; Older Adults; Psychosocial Intervention; Art
MeSH Terms: conditions — Depression; Ageism | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arts group (Experimental): A 9-week Cultural Art Program
  Interventions: Behavioral: Cultural Arts Program
- Waitlist control (Active Comparator): Treatment as usual
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Cultural Arts Program — 9-session group art program using Chinese calligraphy as the channel for gaining emotional awareness and facilitating expression
  Arms: Arts group
Behavioral: Treatment as usual — Treatment as usual provided in local community aged care centres
  Arms: Waitlist control

SUMMARY:
This study examines the effectiveness of an innovative cultural arts program in reducing depressive symptoms and age-related self-stigma among older Chinese as compared to service as usual through a randomized waitlist controlled trial.

DETAILED DESCRIPTION:
Depressive symptoms are common among community-dwelling older people, and prevention and early detection can reduce the incidence of depressive disorders. However, internalized ageism and stigma of mental illness may disempower older people and impede help-seeking behaviors among those at risk of depression. Nonpharmacological interventions may reduce stigma, and among different approaches, arts-based programs are gaining attention because arts are deemed enjoyable, stigma-free, and conducive to mental health.

This study adopts a waitlist-controlled trial and examines the effectiveness of an innovative cultural art programme to combat internalised ageism and reduce depressive symptoms compared with service as usual. Community-dwelling older adults (age 60 years and over) at risk for depression will be recruited and randomised to receive cultural arts (experimental group) or service as usual (waitlist control group). Assessments will be administered by trained researcher(s) at baseline (T0), and completion of the 9-session intervention (T1). Effectiveness analyses will be based on changes in assessments at different time points between intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years or above;
* at risk for depression, i.e., Patient Health Questionnaire (PHQ-9) score under 10; or
* having at least one risk factor of depression, including frequent loneliness, lack of social interaction, lack of meaningful/enjoyable activities, chronic pain, more than four chronic diseases, or bereavement.

Exclusion Criteria:

* known history of autism, intellectual disability, schizophrenia-spectrum disorder, bipolar disorder, Parkinson's disease, or dementia;
* illiterate;
* physically frail; or
* significant suicidal risk.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in depressive symptoms at 9 weeks | Baseline (T0) and 9 weeks after baseline (T1)
  Depressive symptoms are assessed using the Patient Health Questionnaire (PHQ-9) (Kroenke et al., 2001). It is a 9-item instrument that incorporates depression diagnostic criteria with other leading major depressive symptoms and rates the frequency of the symptoms, factoring into the scoring severity index. PHQ-9 scores of 5-9, 10-14, 15-19, 20 and above represent mild, moderate, moderately severe, and severe depression, respectively.
Changes from baseline in self-stigma of age at 9 weeks | Baseline (T0) and 9 weeks after baseline (T1)
  Self-stigma of age is assessed by the Internalized Stigma of old age scale (IS65+) (González-Domínguez et al., 2018). The IS65+ scale is a 9-item instrument comprised of five factors: alienation, discrimination experience, social withdrawal, stigma resistance, and stereotype endorsement. Participants responded to a 4-point Likert scale ranging from 1 (completely disagree) to 4 (completely agree), and a higher score indicates more internalized ageism. The original scale had good internal consistency (α = 0.89).
Changes from baseline in self-stigma of depression at 9 weeks | Baseline (T0) and 9 weeks after baseline (T1)
  Self-stigma of depression is assessed using the 16-item Self-Stigma of Depression Scale (SSDS) (Barney et al., 2006). Questions begin with the stem "If I were depressed, I would …" and include items such as "feel inferior to others" (Shame), "think I should be able to cope with things" (Self-Blame), and "feel I could not contribute much socially" (Social Inadequacy). Participants responded using a 5-point Likert scale of 1 (strongly disagree) to 5 (strongly agree). A higher score indicates more self-stigma of depression, and the scale has good construct validity, internal consistency (α = 0.87) and satisfactory test-retest reliability (Cohen's d = 0.17).

SECONDARY OUTCOMES:
Changes from baseline in empowerment at 9 weeks | Baseline (T0) and 9 weeks after baseline (T1)
  Empowerment is measured by the self-empowerment subscale (SES, four items) from the Mental Health Recovery Measure (MHRM) (Young & Bullock, 2003). Items are rated on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree); higher scores indicate a higher self-reported level of self-empowerment. Example items include: "I believe in myself" and "I have control over my mental health problems"; a higher score indicates more self-empowered.
Changes from baseline in cognitive fusion at 9 weeks | Baseline (T0) and 9 weeks after baseline (T1)
  Cognitive fusion is measured by the self-report Cognitive Fusion Questionnaire (CFQ) (Gillanders et al., 2014). It is a 7-item Likert-type scale ranging from 1 (never true) to 7 (always true). Example items include: "My thoughts cause me distress or emotional pain" and "I tend to get very entangled in my thoughts." Higher scores indicated higher levels of cognitive fusion in participants, ranging from 7 to 49. The scale was validated in Chinese, with good internal consistency (α = 0.92) and test-retest reliability (r = 0.67) (Zhang et al., 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Tianyin Liu, PhD, Principal Investigator — The Polytechnic University of Hong Kong
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT06527625/Prot_SAP_000.pdf